CLINICAL TRIAL: NCT02887781
Title: Clinical Presentation and Renal Outcome of Patients With Tuberous Sclerosis Complex and/or Renal Angiomyolipoma in the Great West Region of France
Acronym: TSAR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: TSAR (RB 14.055)
Record Dates: First submitted 2016-08-30; First posted 2016-09-02 (Estimated); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Tuberous Sclerosis Complex
MeSH Terms: conditions — Tuberous Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood

SUMMARY:
This study aims to investigate the factors (clinical, care-related and genetic) affecting renal outcome in patients with TSC (Tuberous sclerosis complex)

ELIGIBILITY:
Inclusion criteria of study participants

* Patient presenting with an isolated angiomyolipoma or
* Patient presenting with tuberous sclerosis complex combined with an angiomyolipoma or
* Patient presenting with tuberous sclerosis complex
* Patient not objecting to the study

Exclusion criteria of study participants

■Patient objecting to the study

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with TSC and followed in one of the nephrology centers in the West of France
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2015-08-13 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Evolution of the renal function estimated by the MDRD GFR | 18 months after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Yannick LE MEUR, MD PhD, Study Director — University Hospital, Brest
Locations (2):
- France (2):
  - CHU Brest, Brest
  - CHU Rennes, Rennes